CLINICAL TRIAL: NCT04209075
Title: Prebiotics and Metformin Influences Gut and Hormones in Type 2 Diabetes Youth (MIGHTY)
Brief Title: Prebiotics and Metformin Improve Gut and Hormones in Type 2 Diabetes in Youth (MIGHTY-fiber)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 200018; 20-DK-0018 (Other: NIH Clinical Center)
Record Dates: First submitted 2019-12-20; First posted 2019-12-23 (Actual); Results first posted 2022-08-30 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2021-08

CONDITIONS: Diabetes
Keywords: Metformin; Type 2 Diabetes; Youth; Microbiome; Gastrointestinal Side Effects
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo then Prebiotic (Experimental): Participant will take Placebo during Period 1 and Prebiotic during Period 2
  Interventions: Dietary Supplement: Biomebliss; Drug: Metformin; Dietary Supplement: Placebo
- Prebiotic then Placebo (Experimental): Participant will take Prebiotic during Period 1 and Placebo during Period 2
  Interventions: Dietary Supplement: Biomebliss; Drug: Metformin; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Biomebliss — BiomeBliss is a commercially available powder containing prebiotic fiber (inulin and beta glucan), along with blueberry extract providing polyphenols.
Drug: Metformin — Metformin is a commonly used antidiabetic medication, and the only oral medication approved for children and adolescents under 18 years old. Though reasonably effective, gastro-intestinal side effects are common (80% at initiation, and 10-30% after long term use). Metformin dosing at clinically recommended doses will be titrated per protocol during the study.
Dietary Supplement: Placebo — Placebo Comparator

SUMMARY:
Background:

Metformin is a pill youth with type 2 diabetes take. It can cause side effects like diarrhea and upset stomach. Researchers want to see if a fiber supplement can help decrease these side effects.

Objective:

To see if a prebiotic fiber supplement helps improve the gastrointestinal side effects of people taking metformin and helps with their blood sugars.

Eligibility:

People ages 10-25 with type 2 diabetes who are taking or will take metformin

Design:

Participants will be screened with:

Physical exam

Medical history

Blood and urine tests

Meeting with a nutritionist

Participants will stop taking all diabetes medication for 1 week. They will then take metformin by mouth for 1 week. They will be randomly assigned to take either a fiber supplement or a placebo by mouth during the same week. They will then stop all study treatments for 2-3 weeks. Then they will restart metformin for 1 week. The groups that received the fiber versus the placebo will be reversed. All participants will then continue taking metformin and take the fiber for 1 month.

Participants will have 6 visits over about 2 months. These will include:

Blood and urine tests

Meal tests: A plastic tube will be inserted in the participant s arm vein for blood draws. They will drink a special meal.

Dual-energy x-ray absorptiometry (DXA) scan: Participants will lie on their back while the scan measures their body fat and muscle.

While they are home, participants will:

Fill out daily surveys online

Wear daily activity and blood sugar monitors

Collect their stool

Eat only certain foods for two 1-week periods...

DETAILED DESCRIPTION:
Metformin is the most widely prescribed anti-diabetes medication in the world and the first-line therapy for treating type 2 diabetes (T2D) in youth and adults. However, metformin s glucose-lowering ability is variable in clinical practice, and efficacy is further limited by poor medication adherence because of metformin-associated adverse effects. Gastrointestinal (GI) symptoms such as bloating, abdominal discomfort, cramping, and diarrhea are the most common side effects associated with metformin use occurring in up to 80% of individuals at drug initiation and up to 30% in individuals on chronic treatment. In youth with type 2 diabetes, the burden of metformin-associated side effects is high because metformin is the only oral FDA-approved for treatment and there are no other oral alternatives. Therefore, identifying ways to mitigate these GI side effects, especially in youth with type 2 diabetes, is of high clinical significance. New data suggest that metformin-induced changes in the gut and/ or the microbiome may be related to both its beneficial (glucose-lowering) and adverse effects. To address this clinical challenge, prebiotic fibers that are non-digestible food ingredients, may help to improve metformin tolerability by increasing beneficial bacteria and stool metabolites, such as short chain fatty acid (SCFA) stool concentrations. This pilot study will test the hypothesis that a prebiotic microbiome modulator (MM) - containing prebiotic fibers and polyphenols - will reduce GI side effects of metformin at time of initiation and change the stool metabolite profile in youth and young adults with T2D treated with metformin, age 10-25 years who are not on insulin therapy. The 9-week study will have 2 phases and 6 outpatient visits at the NIH Clinical Center. Phase 1 is a 5-week randomized double blind cross-over trial with two 1-week intervention periods (metformin + prebiotic and metformin + placebo) during which subjects will eat a standardized diet. Phase 2 will occur immediately following phase 1 in which participants will start an open-label 4-week intervention with metformin and the prebiotic MM.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age 10-25 years
  2. Pubertal or post-pubertal: Girls - Tanner stage IV-V breast; Boys - Testicular volume >10cc
  3. Diagnosis of type 2 diabetes by American Diabetes Association (ADA) guidelines [36] or with established diagnosis previously treated with metformin.
  4. Negative test for diabetes-related autoantibodies (glutamic acid decarboxylase 65 and tyrosine phosphatase-related islet antigen 2 (IA-2)) documented in NIH CRIS chart or via outside laboratory assessment within the last 10 years.
  5. Hemoglobin A1C <8% at study initiation

EXCLUSION CRITERIA:

1. Pregnancy or breastfeeding
2. Allergy to study medications
3. Allergy or self-reported intolerance to blueberry, pomegranate, or oats, soy, gluten or dairy products.
4. Chronic insulin therapy or insulin use within the last 3 months
5. Treatment with other medications which are known to affect the parameters under study, including antibiotics within the last month, immunosuppressants, proton-pump inhibitors, supraphysiologic systemic steroids, probiotic or prebiotic supplements
6. Heavy yogurt consumption (2 or more servings of >=6 oz per day)
7. Chronic GI disease, gastric bypass surgery, cancer diagnosis or autoimmune disease
8. Metabolic derangement such as metabolic acidosis, severe hyperglycemia (fasting blood glucose >= 200mg/dL), and/or liver enzymes > three times the upper limit of normal.
9. Any other condition that, in the opinion of the investigators, will increase risk to the subject, or impede the

   accurate collection of study-related data.
10. Body weight >= 450lbs
11. Body weight <=58kg
12. Hemoglobin concentration <10g/dL

Ages: 10 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie T Chung, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Burton JH, Johnson M, Johnson J, Hsia DS, Greenway FL, Heiman ML. Addition of a Gastrointestinal Microbiome Modulator to Metformin Improves Metformin Tolerance and Fasting Glucose Levels. J Diabetes Sci Technol. 2015 Jul;9(4):808-14. doi: 10.1177/1932296815577425. Epub 2015 Mar 23. PMID 25802471
- [Derived] Dixon SA, Mishra S, Dietsche KB, Jain S, Mabundo L, Stagliano M, Krenek A, Courville A, Yang S, Turner SA, Meyers AG, Estrada DE, Yadav H, Chung ST. The effects of prebiotics on gastrointestinal side effects of metformin in youth: A pilot randomized control trial in youth-onset type 2 diabetes. Front Endocrinol (Lausanne). 2023 Feb 23;14:1125187. doi: 10.3389/fendo.2023.1125187. eCollection 2023. PMID 36909343
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-DK-0018.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo Then Prebiotic | Prebiotic Then Placebo
Started | 4 | 2
Completed | 4 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Then Prebiotic | Prebiotic Then Placebo | Total
Number analyzed (Participants) | 4 | 2 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 17.5 (0.58) | 16.5 (3.54) | 17.2 (1.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 42.29 (10.9) | 39.41 (2.4) | 41.33 (8.6)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 130.5 (8.3) | 116.5 (17.7) | 125.8 (12.5)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 72.5 (3.0) | 64.5 (3.5) | 69.8 (5.0)

OUTCOME MEASURES:

1. Primary Outcome: Gastrointestinal (GI) Tolerability Score
Description: A composite tolerability score based on 4 GI side effect profile categories (stool consistency, urgency to evacuate, bloating sensation, and flatulence), assessed by daily survey, will be calculated using a principal components analysis. A scale range of GI tolerability score is (1.14, 3.3). A higher tolerability score indicates a lower side effect profile
Time Frame: 1 week (assessed daily for 7 days)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Then Prebiotic | Prebiotic Then Placebo
Number analyzed (Participants) | 4 | 2
score on a scale
  Period 1 | 2.31 (0.62) | 2.63 (0.33)
  Period 2 | 2.70 (0.27) | 2.71 (0.22)

2. Secondary Outcome: Stool Short Chain Fatty Acids (SCFA)
Description: Stool SCFA, including propionate and butyrate, will be measured in stool samples. SCFAs are microbial metabolites that are gut mediators of metabolism.
Time Frame: 1 week and 4 weeks
Population: SCFA analysis of stool samples was not and never will be conducted, data was not collected for this Outcome Measure.
Arm/Group | Placebo Then Prebiotic | Prebiotic Then Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 9 Weeks
Groups:
- Placebo Then Prebiotic: Period 1: Participant will take Placebo during Period 1 and Prebiotic during Period 2
  Biomebliss: BiomeBliss is a commercially available powder containing prebiotic fiber (inulin and beta glucan), along with blueberry extract providing polyphenols.
  Metformin: Metformin is a commonly used antidiabetic medication, and the only oral medication approved for children and adolescents under 18 years old. Though reasonably effective, gastro-intestinal side effects are common (80% at initiation, and 10-30% after long term use). Metformin dosing at clinically recommended doses will be titrated per protocol during the study.
  Placebo: Placebo Comparator
- Prebiotic Then Placebo: Period 1: Participant will take Prebiotic during Period 1 and Placebo during Period 2
  Biomebliss: BiomeBliss is a commercially available powder containing prebiotic fiber (inulin and beta glucan), along with blueberry extract providing polyphenols.
  Metformin: Metformin is a commonly used antidiabetic medication, and the only oral medication approved for children and adolescents under 18 years old. Though reasonably effective, gastro-intestinal side effects are common (80% at initiation, and 10-30% after long term use). Metformin dosing at clinically recommended doses will be titrated per protocol during the study.
  Placebo: Placebo Comparator
- Placebo Then Prebiotic: Period 2: Participant will take Placebo during Period 1 and Prebiotic during Period 2
- Prebiotic Then Placebo: Period 2: Participant will take Prebiotic during Period 1 and Placebo during Period 2
Arm/Group | Placebo Then Prebiotic: Period 1 | Prebiotic Then Placebo: Period 1 | Placebo Then Prebiotic: Period 2 | Prebiotic Then Placebo: Period 2
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/2 | 0/4 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/2 | 0/4 | 0/2
Other Adverse Events (participants affected / at risk) | 1/4 | 0/2 | 4/4 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Then Prebiotic: Period 1 (N=4) | Prebiotic Then Placebo: Period 1 (N=2) | Placebo Then Prebiotic: Period 2 (N=4) | Prebiotic Then Placebo: Period 2 (N=2)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vomitting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoglysemia (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-09): https://cdn.clinicaltrials.gov/large-docs/75/NCT04209075/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-24): https://cdn.clinicaltrials.gov/large-docs/75/NCT04209075/ICF_001.pdf